CLINICAL TRIAL: NCT02531958
Title: Assessment of Optimal Egg Intake in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Maria Luz Fernandez, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H15-227
Record Dates: First submitted 2015-08-20; First posted 2015-08-25 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Eggs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Egg (Experimental): Consumption of 1 egg per day for 4 weeks
  Interventions: Other: Eggs
- 2 Eggs (Experimental): Consumption of 2 eggs per day for 4 weeks
  Interventions: Other: Eggs
- 3 Eggs (Experimental): Consumption of 3 eggs per day for 4 weeks
  Interventions: Other: Eggs

INTERVENTIONS:
Other: Eggs — Participants will complete a 2-week washout period followed by intake of 1, 2, and 3 eggs per day for 4 weeks each.

SUMMARY:
Recently, the United States Department of Agriculture (USDA) has recommended removal of the 300mg/day limit on dietary cholesterol intake due to a lack of evidence supporting a connection between cholesterol intake and increased risk for cardiovascular disease (CVD). Previous work has shown that daily intake of eggs actually favorably alters many parameters associated with CVD risk. Conversely, emerging research suggests that choline, a nutrient in eggs, may be converted into trimethylamine oxide (TMAO) by the intestinal microbiota. TMAO is thought to increase the risk for CVD. Therefore, the purpose of this study is to determine a threshold of daily egg intake at which the risk for CVD is not negatively impacted in a young, healthy population.

DETAILED DESCRIPTION:
The purpose of this study is to establish a threshold of egg intake at which CVD risk is not negatively altered in young, healthy individuals. Participants (age 18-30, healthy lipid profile) will undergo a 2-week washout period followed by daily intake of 1, 2, and 3 eggs per day for 4 weeks each. Blood samples will be collected at baseline and following each 4-week dietary period. Samples will be analyzed to determine the impact of daily intake of increasing numbers of eggs on blood lipids, TMAO, biomarkers of oxidative stress and inflammation, and expression of cholesterol-related genes.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-29.9 kg/m2
* Proficient in English
* Cholesterol ≤ 240 mg/dL
* Willing to consume 1, 2, and 3 eggs per day for 4 weeks each

Exclusion Criteria:

* Diabetes mellitus, cardiovascular disease, history of stroke, renal disease, liver disease, cancer, or eating disorder
* Taking glucose-lowering supplements or medications
* Taking triglyceride-lowering medications, bile acid sequestrants, or high-dose chromium or cinnamon supplements
* Plasma glucose < 126 mg/dL, triglycerides > 500 mg/dL, or blood pressure > 140/90 mmHg (average of 3 readings)
* Allergy to eggs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Plasma high-density lipoprotein (HDL) | 14 Weeks
  Plasma HDL (in mg/dL) will be measured at 2, 6, 10, and 14 weeks to determine the impact of daily egg intake on HDL

SECONDARY OUTCOMES:
Plasma trimethylamine oxide (TMAO) | 14 Weeks
  Plasma levels of TMAO (in µm) will be measured at weeks 2, 6, 10, and 14 to determine the extent to which daily egg intake impacts plasma TMAO concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luz Fernandez, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] DiMarco DM, Norris GH, Millar CL, Blesso CN, Fernandez ML. Intake of up to 3 Eggs per Day Is Associated with Changes in HDL Function and Increased Plasma Antioxidants in Healthy, Young Adults. J Nutr. 2017 Mar;147(3):323-329. doi: 10.3945/jn.116.241877. Epub 2017 Jan 11. PMID 28077734